CLINICAL TRIAL: NCT00970034
Title: Comparative Gene Expression Profiles in Patients With Permanent Atrial Fibrillation and Normal Sinus Rhythm
Brief Title: Gene Expression Profiles in Patients With Permanent Atrial Fibrillation (AF) Versus Sinus Rhythm (SR)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: A. Ruchan Akar, Assoc. Prof., Ankara University
Other Study IDs: 108S375
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Mitral Regurgitation; Atrial Fibrillation; Sinus Rhythm
Keywords: Atrial fibrillation, apoptosis, oligonucleotide microarray
MeSH Terms: conditions — Mitral Valve Insufficiency; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human atrial tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AF: Patients with degenerative mitral valve regurgitation and permanent atrial fibrillation who require mitral valve repair or replacement.
- SR: Patients with degenerative mitral valve regurgitation and maintaining sinus rhythm who require mitral valve repair or replacement.

SUMMARY:
The aim of this project is to determine the morphological criteria of apoptosis in atrial tissues of patients with AF versus SR at transcriptome and genomic size.

DETAILED DESCRIPTION:
Mitral valve regurgitation (MR) is the second most common valvular heart disease encountered in adults. Furthermore, atrial fibrillation (AF) is the most common cardiac arrhythmia seen in clinical practice. Overall, 70% of the patients with severe MR are associated with AF independent from etiopathogenesis of MR. AF is clinically divided into three subgroups; 1) paroxysmal AF, occurs as episodes and ends spontaneously, 2) persistent AF, episodes terminate only with medical or electrical cardioversion, and 3) permanent AF, current medical treatments and electrical cardioversion does not restore a normal sinus rhythm. Despite intensive electrophysiological studies, the molecular mechanisms and pathways of AF are still not fully elucidated.

Apoptosis which has distinctive morphological and biochemical characteristics is genetically regulated, active programmed cell death process. It is known that cardiac morphogenesis restore from apoptosis. In addition, apoptosis has an important role in several cardiovascular system pathologies. It has been shown that atrial apoptosis causes numerous arrhythmias including AF. Likewise, in the pilot study which has been performed by our study group, AF is associated with apoptosis by immunohistochemical and DNA fragmentation analysis methods.

The aim of this project is to determine the morphological criteria of apoptosis in atrial tissues of patients with AF by using electron microscopy and immunohistochemistry. Moreover, we will investigate the transcriptional profile of AF associated genes by oligonucleotide microarray method. The gene expression profiles of patients with AF and degenerative MR will be compared with the atrial tissue samples from the patients with degenerative MR who preserve normal sinus rhythm which will serve as controls. In summary the apoptotic pathways would be analyzed at transcriptomic and genomic level. Besides, the pathways that may interfere AF pathophysiology would also be evaluated. The expression profiles of the genes primarily verified by quantitative real time RT-PCR will be further confirmed by translation of end-result proteins determined with Western blot technique. Thus, brand-new clues about physiology of fibrillating atrial cells would be achieved.

Keywords: Atrial fibrillation, apoptosis, oligonucleotide microarray

ELIGIBILITY:
Inclusion Criteria:

* Patients with permanent atrial fibrillation or sinus rhythm and degenerative mitral valve regurgitation who require cardiac surgery
* Pulmonary hypertension (systolic PA > 45 mmHg)
* Left ventricular ejection fraction > 30%

Exclusion Criteria:

* Paroxysmal AF or atrial flutter
* Second or third degree heart block
* Permanent pacemaker
* Wolff-Parkinson-White syndrome
* Brugada syndrome
* Ischemic or rheumatic mitral valve disease
* Dilated cardiomyopathy
* LVEF < 30%
* Infective endocarditis, myocarditis
* Trauma
* Active HBV, HCV, HIV infection
* Chronic renal failure
* Autoimmune diseases
* Vasculitis
* Known genetic disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Degenerative mitral valve regurgitation who require cardiac valve surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-12; Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Expression profiles of genes related to apoptosis | 6 months

SECONDARY OUTCOMES:
Expression profiles of pro-apoptotic and anti-apoptotic proteins | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: RUCHAN A AKAR, Assoc. Prof., Principal Investigator — Ankara University
Locations (1):
- Ankara University Medical Faculty, Department of Cardiovascular Surgery,, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Cubukcuoglu Deniz G, Durdu S, Dogan Y, Erdemli E, Ozdag H, Akar AR. Molecular Signatures of Human Chronic Atrial Fibrillation in Primary Mitral Regurgitation. Cardiovasc Ther. 2021 Oct 15;2021:5516185. doi: 10.1155/2021/5516185. eCollection 2021. PMID 34737791